CLINICAL TRIAL: NCT05395689
Title: Efficacy and Safety Assessment of a Subcutaneous Immunotherapy (Beltavac®) With Polymerized Allergenic Extract From House Dust Mites in Patients With Allergic Rhinitis/Rhinoconjuntivitis
Brief Title: Efficacy and Safety Assessment of Beltavac® With Polymerized Extract of HDM
Acronym: PROACAROS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Probelte Pharma S.L.U. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-ACAROS-2018-01
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: House Dust Mite Allergy
MeSH Terms: conditions — Dust Mite Allergy | interventions — Antigens, Dermatophagoides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active substance (Experimental): House dust mites allergoid from Dermatophagoides pteronyssinus and Dermatophagoides farinae solution administered by the subcutaneous route for 12 months using a rush schedule
  Interventions: Biological: House dust mites allergoid from Dermatophagoides pteronyssinus and Dermatophagoides farinae
- Placebo (Placebo Comparator): Saline solution administered by the subcutaneous route for 12 months using a rush schedule
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: House dust mites allergoid from Dermatophagoides pteronyssinus and Dermatophagoides farinae — The vaccine will be administered according to a rush schedule meaning one administration each month for 1 year
  Arms: Active substance
Biological: Placebo — The vaccine will be administered according to a rush schedule meaning one administration each month for 1 year
  Arms: Placebo

SUMMARY:
The trial is performed to assess efficacy and safety of Beltavac with polymerized extract of house dust mites in allergic Rhinoconjunctivitis associated or not with asthma

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, signed and duly dated.
* Man or woman between 12 and 65 years old (both included).
* Patient with moderate or severe symptoms of persistent rhinitis according to the ARIA Guide, associated or not with well or partially controlled asthma according to the GEMA 5.0 Guide.
* Confirmation of sensitization to DPT or DF with a positive prick test (mean papule diameter greater than or equal to 3 mm) with a commercial standardized allergenic extract and a serum extract-specific IgE value of class 3 or higher (> 3.5 kU / L) within the 6 months prior to the study.
* Negative pregnancy test.
* Nasal symptom and medication combined scale score ≥ 1.5 during the screening phase.

Exclusion Criteria:

* Concomitant sensitization to allergens other than dust mites if clinically relevant symptoms are anticipated that may interfere with study evaluation periods at the discretion of the investigator.
* Poorly controlled asthma according to the GEMA 5.0 guideline
* Severe asthma, that is, those who during the last months have controlled their asthma according to therapeutic step 5-6 of the GEMA 5.0 guideline.
* Autoimmune diseases or immunodeficiency.
* Malignant neoplasms, serious cardiovascular disease, serious mental illness or other relevant chronic diseases that may interfere with the results of the study.
* Clinical history of anaphylaxis with cardio / respiratory symptoms.
* Hypersensitivity to any of the excipients of the investigational product.
* Immunosuppressive medication during the last 6 months before the inclusion of patients and until the end of the study.
* Treatment with beta-blockers during the study.
* Patients who have previously received immunotherapy with allergenic dust mite extract or other extracts and have failed within the last 5 years.
* Patients with immunotherapy with allergens other than dust mites during the study period.
* Patients who receive any other vaccine one week before the start of treatment or awaiting the second dose of vaccine against COVID-19.
* Pregnant or nursing patients.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The combined nasal symptom and medication score | 12 months of treatment
  The symptoms assessed are: itchy nose, sneezing, runny nose, and blocked nose (all rated from 0-3). The medication score is 1 for oral and/or topical antihistamines, 2 for intranasal corticosteroids, and 3 for oral corticosteroids. The scores from the nasal symptoms are added and divided by 4 to a total daily symptom score from 0-3.Final score range from 0 to 6, higher score meaning a worse outcome.

SECONDARY OUTCOMES:
Score of the nasal symptoms scale | 12 months of treatment
  Symptoms assessed are: itchy nose, sneezing, runny nose, and blocked nose (all rated from 0-3). Final score range from 0 to 3, higher score meaning worse outcome.
Score of the specific medication scale | 12 months of treatment.
  The medication score is 1 for oral and/or topical antihistamines, 2 for intranasal corticosteroids, and 3 for oral corticosteroids. Final score range from 0 to 3, higher score meaning worse outcome.
Percentage of days without symptoms or medication | 12 months of treatment
  Percentage of days with a zero value for symptom and medication recorded in the patient digital diary
VAS score (completed by the patient and the investigator) | 12 months of treatment.
  Visual analogue score from 0 (no symptoms) to 100mm (serious symptoms) to assess global symptoms of allergy
RCAT questionnaire | 12 months of treatment.
  Rhinitis Control Assessment Test. Score from 6 (poor control) to 30 (good control)
Mini-RQLQ questionnaires | 12 months of treatment.
  Mini-Rhinoconjunctivitis Quality of Life Questionnaire
Values in serum of specific IgE and IgG4 | 12 months of treatment.
  Specific IgE and IgG4 to DPT and total DF, Der p1 and Der p2, Der p23, Der f1, Der f2
Number of local and systemic reactions. | 13 months of study follow up
  Number of local and systemic reaccions associated with the treatment
Cost-effectiveness analysis | 13 months of study follow up
  Number days/ visits related to allergy
The combined asthma symptom and medication score | 12 months of treatment
  The symptoms assessed are: symptoms during the day, symptoms during the night and physical activity limitations (all rated from 0-3). The medication score is 1 for inhalated corticoids (low dose) , 2 for inhalated corticosteroids associated with LABA, and 3 for inhalated corticosteroids medium dosis associated with LABA. The scores from the symptoms are added and divided by 3 to a total daily symptom score from 0-3. The total daily medication score ranges from 0-3.
PEF | 12 months of treatment
  Peak expiratory flow measured with a Smart Peak Flow device
ACT questionnaire | 12 months of treatment
  Asthma Control Test Questionnaire to assess the control of asthma in asthmatic patients

CONTACTS AND LOCATIONS:
Locations (18):
- Spain (18):
  - Hospital Vega Baja, Orihuela, Alicante
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital de la Plana, Castellon, Castellón
  - Hospital Regional de Málaga, Málaga, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Fundacion Sanitaria Sant Pere Claver, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital infantil Vall d Hebron, Barcelona
  - Hospital Val d ' Hebron, Barcelona
  - Hospital General de Castellón, Castelló
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital de Fatima, Seville
  - Hospital Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Politecnico de la Fé, Valencia
  - Hospital Universitario Infantil de la Fé, Valencia

IPD SHARING:
Plan to Share IPD: No